CLINICAL TRIAL: NCT06467097
Title: A Phase Ⅲ Randomized Study Systemic Treatment Alone Versus Systemic Treatment Plus Stereotactic Abative Body Radiotherapy for Patients With Oligometastatic Renal Cell Carcinoma: SABLOR Study
Brief Title: Systemic Treatment Alone Versus Systemic Treatment Plus Radiotherapy in Oligometastatic Renal Cell Carcinoma
Acronym: SABLOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Park, Won Park, M.D., Ph.D., Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2023-04-044
Record Dates: First submitted 2024-06-11; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Kidney Neoplasm
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: 1. Control group: A group that undergoes standard treatment alone for metastatic renal cell carcinoma.
  2. Experimental group: A group that receives concurrent radiotherapy for all metastatic lesions in addition to standard treatment.
  We will compare the one-year progression-free survival rate between these groups, randomized from a random allocation point. Block randomization will be used, with 44 participants randomly assigned to each group using a random number table generated from a web-based program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (No Intervention): Only standard treatment is administered. The standard treatment includes targeted cancer therapy, immunotherapy, or monotherapy with each therapeutic agent.
- B group (Experimental): This group receives concurrent partial nephrectomy radiotherapy for all metastatic lesions in addition to standard treatment.
  Interventions: Radiation: SBRT(Stereotatic Body Radiation Therapy)

INTERVENTIONS:
Radiation: SBRT(Stereotatic Body Radiation Therapy) — Patients will receive treatment for one to two weeks, one to five times per region.
  Arms: B group

SUMMARY:
To evaluate whether incorporating locoregional radiotherapy in the treatment of oligometastatic renal cell carcinoma, including inductive oligometastases, along with standard systemic therapy, contributes to improved progression-free survival rates for patients.

DETAILED DESCRIPTION:
Various institutions are attempting to use locoregional radiotherapy in the treatment of oligometastatic renal cell carcinoma, accompanied by a few metastases. Research findings have indicated that high-dose locoregional radiotherapy can suppress disease progression, potentially prolonging the interval for additional systemic therapy; however, whether the addition of locoregional radiotherapy in cases of renal cell carcinoma with oligometastases demonstrates superior oncologic outcome compared to standard systemic therapy alone has yet to be established. Therefore, a randomized phase III study is being conducted to evaluate whether incorporating locoregional radiotherapy in the treatment of oligometastatic renal cell carcinoma, including inductive oligometastases, along with standard systemic therapy, contributes to improved progression-free survival rates for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic renal cell carcinoma classified within the ESTRO/EORTC classification system as having ≤ 5 metastases, ≤ 3 metastatic organs, and meeting criteria for new, recurrent, or induced metastases.
2. Patients aged 20 to 80 years.
3. Patients with individual metastases ≤ 5 cm in longest diameter.
4. Patients with primary tumors surgically removed or scheduled for surgery.
5. Patients histologically diagnosed with clear cell carcinoma.
6. Patients with ECOG performance status 0-1.
7. Patients with normal major organ function and bone marrow function meeting specific criteria: WBC ≥ 2,000/μL, neutrophils ≥ 1,000/μL, platelets ≥ 50,000/μL.
8. Patients who understand the contents of the informed consent form, voluntarily consent to participate in the study, and sign the informed consent form.
9. Patients who agree to use contraception from the time of signing the consent form until 1 year after the last standard systemic therapy.
10. Breastfeeding women who agree to stop breastfeeding for at least 5 months after the last standard systemic therapy.
11. Patients with visible tumors outside the scope of tumor removal surgery (surgical therapy) for metastatic lesions.

Exclusion Criteria:

1. Patients with total bilirubin > 3.6 mg/dL.
2. Patients with AST >160 U/L, ALT > 165 U/L.
3. Patients unable to maintain position for partial nephrectomy radiotherapy.
4. Patients with a history of radiotherapy to metastatic renal cell carcinoma or surrounding areas.
5. Patients with confirmed brain, peritoneal, or pleural metastases.
6. Patients diagnosed with another solid tumor and treated within 2 years or with residual lesions.
7. Patients who do not consent to participate in the study.
8. Pregnant patients.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2031-02-13 (Estimated); Study Completion 2031-02-13 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival rate | One year after completion of enrollment
  Compare free survival between the standard systemic therapy alone group and systemic therapy combined with radiotherapy group

SECONDARY OUTCOMES:
Local control rate for radiation therapy site at one year | One year after radiation completion of each participant
  Compare Local control rate between the standard systemic therapy alone group and systemic therapy combined with radiotherapy group
Grade 3 acute adverse event | three to six months after study treatment
  Compare acute adverse events according to CTCAE V5.0 between the standard systemic therapy alone group and systemic therapy combined with radiotherapy group
Grade 3 chronic adverse event | one year to three years after radiation completion
  Compare chronic adverse events according to CTCAE V5.0 between the standard systemic therapy alone group and systemic therapy combined with radiotherapy group
Overall survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Compare Overall survival rate between the standard systemic therapy alone group and systemic therapy combined with radiotherapy group

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No